CLINICAL TRIAL: NCT06950671
Title: Role of TREM-1 as a Novel Biomarker in HER-2 Negative Breast Cancer: a Molecular and Clinical Study
Brief Title: Role of Triggering Receptor Expressed on Myeloid Cells (TREM-1) as a Novel Biomarker in Human Epidermal Growth Factor Receptor -2 (HER-2) Negative Breast Cancer: a Molecular and Clinical Study
Status: Not yet recruiting | Type: Observational
Sponsor: Rahma Esam Salama Esawi (Other)
Collaborators: Assiut University (Other)
Responsible Party: Sponsor-Investigator, Rahma Esam Salama Esawi, Role of TREM-1 as a novel biomarker in HER-2 breast cancer : a molecular and clinical study, Assiut University
Organization: Assiut University (Other)
Other Study IDs: novel biomarker in cancer
Record Dates: First submitted 2025-04-19; First posted 2025-04-30 (Actual); Last update posted 2025-04-30 (Actual); Status verified 2025-04

CONDITIONS: Breast Cancer Stage I; Breast Cancer Stage II; Breast Cancer Stage III; Breast Cancer Invasive
Keywords: TREM-1 in non metastatic HER-2 negative breast cancer
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — blood sample will be analyzed by flowctometry
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
Global cancer statistics by world region for the year 2022 estimated breast cancer the 2nd cause of new cancer cases (11.6%). (1) Approximately 80% of all breast cancers (BCs) are currently categorized as human epidermal growth factor receptor 2 (HER2)-negative. (2) Most breast cancer cases can be cured by multimodality treatment, although cure rates vary by clinical stage, subtype and the clinical behavior of cancer which affected by the composition of pro- and anti-tumor immune mediators within the tumor microenvironment. (3, 4) Immune gene signatures in breast tumors -that comprise genes with specialized roles in immune biology- Significantly, have been shown to correlate with patient survival outcomes. (5-8)chemotherapy responsiveness. (7, 9), and more recently, response to immunotherapies.(10-12)One such candidate, the gene encoding Triggering Receptor Expressed on Myeloid Cells (TREM)-1, which emerged as a robust therapy predictive and prognostic marker. TREM1 encodes a type I trans-membrane receptor of the Ig superfamily expressed by effectors of innate immunity including neutrophils, monocytes and macrophages. The TREM-1 receptor is known to augment inflammatory signaling in response to infectious pathogens by promoting release of cytokines that modulate the activation, recruitment and survival of myeloid and lymphoid cells. (13) In this study we hope to gain a better understanding of TREM-1 clinical and molecular relevance in HER2 negative BC either triple negative or hormonal positive which represent significant subset that lack target therapeutic options, evaluating its effect as predictive and prognostic marker and so the potential implications for patient management.

DETAILED DESCRIPTION:
a prospective observational cohort study on the role of TREM-1 as a novel immune biomarker in HER-2 breast cancer it's a molecular and clinical study. our aim is to assess prognostic significance of TREM-1 expression at baseline and post neo-adjuvant treatment regards DFS & OS and to quantify TREM-1 expression and correlate its level with clinical and pathological response to neo-adjuvant treatment. and evaluate its association with immune cells (eg. monocytes and neutrophils)

ELIGIBILITY:
Inclusion Criteria:

* female patient aged < 18 yrs. old
* histological proven breast cancer
* HER-2 negative (hormonal positive or triple negative)
* planned to receive neo-adjuvant therapy
* complete clinical, radiological and therapeutic data

Exclusion Criteria:

* metastatic breast cancer
* HER-2 positive
* incomplete clinical, radiological or therapeutic data

Ages: 18 Years to 80 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — females
Study Population: female patients with HER-2 breast cancer not metastatic planned to receive neoadjuvant therapy
Sampling Method: Probability Sample
Enrollment: 1 (Estimated)
Dates: Start 2025-09-15 (Estimated); Primary Completion 2028-09-15 (Estimated); Study Completion 2029-09 (Estimated)

PRIMARY OUTCOMES:
: assess prognostic significance of TREM-1 expression at baseline and post neo-adjuvant treatment regards DFS & OS | follow up patients over 2 years
  prognostic significance of TREM-1 expression at baseline and post neo-adjuvant treatment regards DFS & OS

CONTACTS AND LOCATIONS:
Overall Officials: summar mohamed summar el-morshidy, lecturer, Study Director — Assiut University
Locations (1):
- Assiut University Hospitals, Asyut, Egypt, Egypt

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Pullikuth AK, Routh ED, Zimmerman KD, Chifman J, Chou JW, Soike MH, Jin G, Su J, Song Q, Black MA, Print C, Bedognetti D, Howard-McNatt M, O'Neill SS, Thomas A, Langefeld CD, Sigalov AB, Lu Y, Miller LD. Bulk and Single-Cell Profiling of Breast Tumors Identifies TREM-1 as a Dominant Immune Suppressive Marker Associated With Poor Outcomes. Front Oncol. 2021 Dec 8;11:734959. doi: 10.3389/fonc.2021.734959. eCollection 2021. PMID 34956864
- See also: Related Info — https://pubmed.ncbi.nlm.nih.gov/34956864/